CLINICAL TRIAL: NCT06977347
Title: Verification of Anti-pseudomonal Antibiotic Combination Therapy in Severe Community-acquired Pneumonia in South Korea: A Randomized-controlled Study
Brief Title: Appropriateness of Antibiotic Combination Therapy for Severe Community-acquired Pneumonia in South Korea
Acronym: ACTSCAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHOSEOK YOON (Other)
Responsible Party: Sponsor-Investigator, CHOSEOK YOON, Clinical Professor, Division of Infectious Diseases, Department of Internal Medicine, Hanyang University Hospital, Seoul, South Korea, Seoul Hospital
Organization: Seoul Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYUH 2025-02-033-002
Record Dates: First submitted 2025-05-09; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Severe Community-acquired Pneumonia (sCAP)
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Piperacillin, Tazobactam Drug Combination; Piperacillin; Tazobactam; Levofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piperacillin/Tazobactam Monotherapy (Experimental): Patients receive empirical treatment with piperacillin/tazobactam alone for severe community-acquired pneumonia. The antibiotic is administered according to standard dosing guidelines for hospitalized patients.
  Interventions: Drug: Piperacillin/Tazobactam
- Piperacillin/Tazobactam Plus Levofloxacin Combination Therapy (Active Comparator): Patients receive empirical combination treatment with piperacillin/tazobactam and levofloxacin for severe community-acquired pneumonia. Both antibiotics are administered concurrently according to institutional protocols for combination therapy.
  Interventions: Drug: Piperacillin/tazobactam + Levofloxacin

INTERVENTIONS:
Drug: Piperacillin/Tazobactam — Piperacillin/tazobactam: 4.5g IV q6h (over 3h)
  Arms: Piperacillin/Tazobactam Monotherapy
Drug: Piperacillin/tazobactam + Levofloxacin — Piperacillin/tazobactam: 4.5g IV q6h (over 3h)
  + Levofloxacin 750mg IV q24h (over 30min)
  Arms: Piperacillin/Tazobactam Plus Levofloxacin Combination Therapy

SUMMARY:
This study aims to provide high-level evidence for appropriate empirical antibiotic use tailored to the clinical reality in Korea by conducting a randomized controlled trial comparing monotherapy with piperacillin/tazobactam and combination therapy with piperacillin/tazobactam plus a fluoroquinolone in patients with severe community-acquired pneumonia.

ELIGIBILITY:
* Inclusion Criteria:

  * Adult patients aged 19 years or older who visited the emergency department and were hospitalized.
  * Findings consistent with pneumonia diagnosis, meeting all of the following criteria:
  * Radiologic evidence of pulmonary infiltration on chest X-ray or chest CT.
  * At least two or more of the following clinical signs:

    i) Body temperature ≥38°C or <36°C ii) White blood cell count ≥11,000/µL or <4,000/µL iii) Presence of purulent sputum or bronchial secretions
  * Within 24 hours of admission, the patient meets one major criterion or three minor criteria according to ATS/IDSA classification:

    * Major criteria:

      i) Invasive mechanical ventilation ii) Use of vasopressors (vasopressor-dependent septic shock)
    * Minor criteria:

      i) Respiratory rate ≥30 breaths/min ii) PaO2/FiO2 ≤ 250 iii) Multilobar infiltrates iv) Confusion or disorientation v) BUN ≥20 mg/dL vi) WBC <4,000/mm³ vii) Platelet count <100,000/mm³ viii) Hypothermia (temperature <36°C) ix) Hypotension requiring aggressive fluid resuscitation
* Exclusion Criteria:

  * Transferred from another hospital after >48 hours of hospitalization
  * Died within 72 hours of hospital admission
  * Transferred to another hospital within 14 days of admission
  * Pneumonia occurring after >48 hours of mechanical ventilation, including home ventilators
  * Detection of influenza or SARS-CoV-2 virus within 7 days of hospitalization
  * Identified non-pneumonia infection requiring antibiotics within 72 hours of admission
  * Detection of piperacillin/tazobactam-resistant Enterobacterales, Pseudomonas spp., or Acinetobacter spp. in respiratory or blood cultures within the past 90 days
  * Antibiotic-related adverse events observed within 72 hours of assigned treatment, requiring discontinuation or change of antibiotics

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
All-cause 28-day mortality | 28 days
  Mortality from any cause within 28 days of randomization.

SECONDARY OUTCOMES:
Need for mechanical ventilation | Up to hospital discharge or 28 days, whichever comes first
  Proportion of patients requiring invasive mechanical ventilation during hospitalization.
ICU admission rate | Up to hospital discharge or 28 days, whichever comes first
  Proportion of patients who require admission to the intensive care unit (ICU) during hospitalization
Length of hospital stay | Up to hospital discharge or 28 days, whichever comes first
  Total number of days from admission to discharge
Time to fever resolution | Up to 7 days after treatment initiation
  Time in days from initiation of antibiotic treatment to the first documented temperature < 37.8°C maintained for at least 24 hours without antipyretic use
Antibiotic-related adverse events | From first dose to 28 days post-treatment
  Incidence of adverse drug reactions associated with study antibiotics (e.g., gastrointestinal symptoms, allergic reactions, hepatotoxicity, nephrotoxicity) as assessed by the treating physician
14-day hospital readmission rate | 14 days after end of antibiotic treatment
  Proportion of patients who are readmitted to any hospital for any cause within 14 days after completion of antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding patient confidentiality and data protection, as well as the lack of a data-sharing infrastructure or formal data request mechanism at this time.